CLINICAL TRIAL: NCT01212315
Title: Triclosan-coated Sutures in Cardiac Surgery:Effects on Leg Wound Infections and Costs
Brief Title: Effects of Triclosan-coated Sutures in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Jeppssons, Professor, Cardiothoracic surgery, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Postoperative Wound Infection
Keywords: Wound infection; SSI; Suture
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Ordinary sutures (Vicryl / Monocryl) is used for wound closure
- Group A (Active Comparator): Triclosan coated sutures (Vicryl Plus / Monocryl Plus) is used for wound closure
  Interventions: Device: Triclosan coated sutures

INTERVENTIONS:
Device: Triclosan coated sutures — Subcutaneous and cutaneous sutures coated with triclosan (Vicryl Plus / Monocryl Plus) are used to close the incisions after vein harvesting and sternotomy. All wounds are inspected before discharge from hospital and the patients are instructed to contact the study coordinator if any suspected infection occurs. In addition, all patients are controlled after thirty days by a nurse and contacted by telephone sixty days after surgery to assess postoperative infections by a predefined questionnaire. Infection symptoms are graded according to the Asepsis score and the CDC classification. Patient records including bacterial cultures and antibiotic treatment are collected for all patients with suspected infections.
  Other Names: Monocryl Plus suture; Vicryl Plus suture
  Arms: Group A

SUMMARY:
The purpose of this study is to assess if triclosan-coated sutures reduces wound infections after saphenous vein harvesting in CABG patients. Secondary objectives are the effect triclosan-coated sutures on sternal wound infections and a cost analysis.

DETAILED DESCRIPTION:
The role of the suture material for the development of postoperative wound infection has been debated for many years. It has been reported that fewer bacteria adhere to monofilament polypropylene than braided polyester sutures in vitro but the results are opposed by a non-randomized clinical study where the use of monofilament sutures was identified as an independent risk factor for leg wound infections after CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective CABG at Sahlgrenska University Hospital with intended use of saphenous vein graft are included.

Exclusion Criteria:

* Patients with on-going sepsis or septicaemia, bacterial infections or known allergy to triclosan are excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with leg wound infection. | Within 60 days after heartsurgery
  Primary endpoint is postoperative leg wound infection within 60 days after surgery according to the definition of Center for Disease Control.

SECONDARY OUTCOMES:
Culture-proven and antibiotic-treated wound infection after heart surgery | Within 60 days after heart surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jeppsson, MD PhD, Principal Investigator — Sahlgrenska Univerity Hospital
Locations (1):
- Dep of Cardiovascular Surgery and Anesthesia, Sahlgrenska Univerity Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Steingrimsson S, Thimour-Bergstrom L, Roman-Emanuel C, Schersten H, Friberg O, Gudbjartsson T, Jeppsson A. Triclosan-coated sutures and sternal wound infections: a prospective randomized clinical trial. Eur J Clin Microbiol Infect Dis. 2015 Dec;34(12):2331-8. doi: 10.1007/s10096-015-2485-8. Epub 2015 Oct 2. PMID 26432552
- [Derived] Thimour-Bergstrom L, Roman-Emanuel C, Schersten H, Friberg O, Gudbjartsson T, Jeppsson A. Triclosan-coated sutures reduce surgical site infection after open vein harvesting in coronary artery bypass grafting patients: a randomized controlled trial. Eur J Cardiothorac Surg. 2013 Nov;44(5):931-8. doi: 10.1093/ejcts/ezt063. Epub 2013 Feb 22. PMID 23435526